CLINICAL TRIAL: NCT00034294
Title: A Randomized, Double-Blind Study of GT160-246 Versus Vancomycin in Patients With C. Difficile-Associated Diarrhea
Brief Title: A Study of GT160-246 Versus Vancomycin in Patients With Clostridium Difficile-Associated Diarrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GTC-80-203; GT1105
Record Dates: First submitted 2002-04-24; First posted 2002-04-25 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Clostridium Difficile-Associated Diarrhea; Clostridium Enterocolitis; Clostridium Difficile Diarrhea; Antibiotic-associated Colitis; Antibiotic-associated Diarrhea
Keywords: C. difficile-associated diarrhea; CDAD; Clostridium difficile-Associated Diarrhea; Clostridium enterocolitis; antibiotic-associated diarrhea; clostridium difficile colitis; infectious diarrhea; chronic diarrhea; antibiotic-associated colitis
MeSH Terms: conditions — Enterocolitis, Pseudomembranous; Dysentery | interventions — styrenesulfonic acid polymer

INTERVENTIONS:
Drug: GT160-246

SUMMARY:
Approximately 300 patients will be entered into this study taking place throughout the United States, Canada and the United Kingdom. This study aims to determine if an investigational drug is safe and effective for treating the symptoms of C. difficile-associated diarrhea and lowering the risk of repeat episodes of diarrhea. The investigational drug will be evaluated in comparison to current standard antibiotic treatment, so all patients will receive active medication.

All study-related care is provided including doctor visits, physical exams, laboratory tests and study medication. Total length of participation is approximately 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old.
* Have active mild to moderate C. difficile- Associated Diarrhea (CDAD).
* Be able to tolerate oral medication.
* Not be pregnant or breast-feeding.
* Sign and date an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-02; Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (88):
- United States (53):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Sacramento, California
  - Newark, Delaware
  - Bay Pines, Florida
  - Brandon, Florida
  - Hollywood, Florida
  - Naples, Florida
  - Orlando, Florida
  - Austell, Georgia
  - Columbus, Georgia
  - Chicago, Illinois
  - Maywood, Illinois
  - North Chicago, Illinois
  - Columbus, Indiana
  - Des Moines, Iowa
  - Wichita, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Chevy Chase, Maryland
  - Boston, Massachusetts
  - Braintree, Massachusetts
  - West Roxbury, Massachusetts
  - Springfield, Missouri
  - St Louis, Missouri
  - Stratford, New Jersey
  - Buffalo, New York
  - Jamaica, New York
  - Manhasset, New York
  - New York, New York
  - Syracuse, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Fargo, North Dakota
  - Columbus, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Allentown, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Upland, Pennsylvania
  - Charleston, South Carolina
  - Clarksville, Tennessee
  - Memphis, Tennessee
  - Temple, Texas
  - Falls Church, Virginia
  - Richmond, Virginia
  - Seattle, Washington
- Canada (10):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Moncton, New Brunswick
  - Ottawa, Ontario
  - Windsor, Ontario
  - Chicoutimi, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Trois-Rivières, Quebec
- Hato Rey, Puerto Rico
- United Kingdom (24):
  - Heathpark, Cardiff
  - Penlan Rd, Cardiff
  - Steeton, Keighley
  - Bury, Lancashire
  - Chelsea, London
  - South Kensington, London
  - High Heaton, Newcastle-upon-Tyne
  - Cliftonville, Northampton
  - Fulwood, Preston
  - Livilands, Stirling
  - Morriston, Swansea
  - Birmingham
  - Cambridge
  - Edinburgh
  - Glasgow
  - Hull
  - Leeds
  - Leicester
  - London
  - Newport
  - Nottingham
  - Shrewsbury
  - Taunton
  - Wolverhampton